CLINICAL TRIAL: NCT03378973
Title: The Effects of Dexmedetomidine Dose on Motor Evoked Potentials During Spine Surgery: A Randomized, Single-blind Trial
Brief Title: The Effects of Dexmedetomidine Dose on Motor Evoked Potentials
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No longer clinically relevant
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017-1304
Record Dates: First submitted 2017-12-12; First posted 2017-12-20 (Actual); Results first posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Spinal Fusion
Keywords: motor evoked potentials
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The anesthesiologist administering anesthetic agents will have knowledge of their doses. The technologist performing motor evoked potential testing and other participants will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High dose dexmedetomidine (Experimental): Patients will receive dexmedetomidine 0.5 mcg/kg/hr plus propofol 50 mcg/kg/min
  Interventions: Drug: Dexmedetomidine
- Low dose dexmedetomidine (Active Comparator): Patients will receive dexmedetomidine 1.0 mcg/kg/hr plus propofol 25 mcg/kg/min
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will randomly assigned to received Arm 1 anesthesia or Arm 2 anesthesia during surgery.
  Other Names: Precedex

SUMMARY:
This a parallel group, two-arm, randomized superiority trial that will compare the effect of two different doses of dexmedetomidine on motor evoked potentials during spine surgery

DETAILED DESCRIPTION:
This a parallel group, two-arm, randomized superiority trial that will compare the effect of two different doses of dexmedetomidine on suitability of motor evoked potentials for intraoperative monitoring during spine surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing multi-level posterior spine fusions requiring motor evoked potential monitoring

Exclusion Criteria:

* Allergy to dexmedetomidine, propofol
* Conditions knows to make recording of motor evoked potentials difficult, including poorly controlled diabetes, severe peripheral neuropathy, severe myelopathy, or previous surgery during which motor evoked potentials were difficult to obtain
* Hepatic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Emerson, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Dexmedetomidine: Patients will receive dexmedetomidine 0.5 mcg/kg/hr plus propofol 50 mcg/kg/min
  Dexmedetomidine: Patients will randomly assigned to received Arm 1 anesthesia or Arm 2 anesthesia during surgery.
- Highdose Dexmedetomidine: Patients will receive dexmedetomidine 1.0 mcg/kg/hr plus propofol 25 mcg/kg/min
  Dexmedetomidine: Patients will randomly assigned to received Arm 1 anesthesia or Arm 2 anesthesia during surgery.
Period: Overall Study
Arm/Group | Low Dose Dexmedetomidine | Highdose Dexmedetomidine
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Dexmedetomidine | Low Dose Dexmedetomidine | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (29) | 53 (21) | 53 (22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Monitorable of Motor Evoked Potentials
Description: Monitorable is defined as stable signals being present in 3 muscles in each lower extremity, with mean peak-to-peak amplitude of at least 50 uV, and with mean-normalized interquartile variability of 0.9 or less.
Time Frame: During a single surgery for the duration of the operation
Measure: Count of Participants; unit: Participants
Groups:
- High Dose Dexmedetomidine: Patients will receive dexmedetomidine 1.0 mcg/kg/hr plus propofol 25 mcg/kg/min
  Dexmedetomidine: Patients will randomly assigned to received Arm 1 anesthesia or Arm 2 anesthesia during surgery.
Arm/Group | Low Dose Dexmedetomidine | High Dose Dexmedetomidine
Number analyzed (Participants) | 4 | 3
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: From time of consent through the duration of surgery
Arm/Group | Low Dose Dexmedetomidine | High Dose Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT03378973/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT03378973/Prot_SAP_002.pdf